CLINICAL TRIAL: NCT00998673
Title: Randomized Standard-of-Care-Controlled Trial of a Silica Gel Fiber (SGF) Wound Dressing in the Treatment of Chronic Venous Leg Ulcers
Brief Title: Silica Gel Fiber Wound Dressing for Chronic Venous Leg Ulcers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGF271-01
Record Dates: First submitted 2009-10-02; First posted 2009-10-20 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Venous Ulcer
Keywords: Silica gel fiber; Chronic venous leg ulcers; Venous ulcer; Stasis ulcer; Varicose ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Device: Silica Gel Fiber
- Arm 2 (Other)
  Interventions: Device: Standard-of-Care

INTERVENTIONS:
Device: Silica Gel Fiber — Silica Gel Fiber (SGF) applications as required
  Arms: Arm 1
Device: Standard-of-Care — Standard-of-Care with dressing changes twice per week using Mepitel and Mepilex wound dressings
  Arms: Arm 2

SUMMARY:
Silica Gel Fiber is a bioresorbable, inorganic silica gel fibre patch promoting skin tissue growth and enhanced wound healing for all types of chronic wounds. It is applied as patch and will be hold in place by a secondary dressing for maintaining the moist wound environment. The study is aimed to demonstrate superiority over a standard wound treatment for chronic venous leg ulcers. The primary efficacy variable is time to healing.

ELIGIBILITY:
Inclusion Criteria:

* At least one chronic venous leg ulcer fulfilling all of the following criteria:

  * Size: >/= 5 cm2 and </= 40 cm2 (measured by Visitrak Wound Measurement System)
  * Duration: >/= 3 month < 5 years
  * Location: Between and including knee and ankle
  * Depth: Involving dermis, with no exposed muscle, tendon or bone. Characterized by a viable wound bed with granulation tissue
  * The etiology of the ulcer as "venous" is proven by Duplex or Doppler sonography and with ankle/brachial arterial Doppler pressure index > 0.8 (exclusion criterion for peripheral arterial disease) and < 1.3 (exclusion criterion for medial sclerosis), or with a laser Doppler value > 40
* Treatment with active wound care agents paused for 14 days before start of study treatment

Exclusion Criteria:

* Only ulcers of other than venous etiology, e.g., diabetic ulcers or ulcers resulting from electrical, chemical, or radiation insult, after contact eczema, etc.
* History of radiotherapy to the target ulcer site
* Signs of infection as defined by rubor, dolor, calor, tumor, functio laesa. Fever (38°C sublingual, rectal, or ear), rigors, or leukocytosis will be considered as signs of infection in the context of the general appearance of the wound
* Target ulcer lacking any sign of granulation tissue (bradytrophic wound bed)
* Presence of necrotic tissue
* Presence of fistula
* History of connective tissue disease, e.g., systemic lupus erythematodes, systemic sclerosis, Sjögren's syndrome or mixed connective tissue disease
* Uncontrolled congestive heart failure
* Malnutrition (albumin < 2.5 g/dl; to be measured if clinical signs of malnutrition are being observed)
* Uncontrolled diabetes (HbA1c > 8 %)
* Previous organ transplantation
* Active malignant disease
* Severe rheumatoid arthritis
* Undergoing haemodialysis
* Active sickle cell disease
* Patients who are immunocompromised for reasons such as therapy with corticosteroids, chemotherapy, antiangiogenic or immunosuppressive agents, or due to immunodeficiency syndromes
* Pregnant or nursing women
* Woman of childbearing potential who are not practicing acceptable methods of birth control during the investigation period
* Known allergy to any of the devices' constituents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Time to healing of target ulcer, defined as the treatment period day during the weekly visit at which the surface area of the wound was noted as zero and completely healed | Week 12

SECONDARY OUTCOMES:
Incidence of complete wound healing of target ulcer at 4, 8 and 12 weeks, defined as full epithelialisation of the wound with the absence of drainage | Week 4/8/12
Rate of recurrence of wound at end of follow-up period of 3 months | Week 24
Size (cm2, measured by Visitrak Wound Measurement System) of target ulcer (Absolute size measured once per week and change between assessments at weeks 0, 4, 8, and 12) | Week 12/24

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- Germany (14):
  - Berlin
  - Bochum
  - Bonn
  - Cologne
  - Dresden
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Göttingen
  - Greifswald
  - Hamburg
  - Mannheim
  - Regensburg
  - Ulm